CLINICAL TRIAL: NCT02393755
Title: A Phase I/II Study of Nintedanib and Capecitabine in Refractory Metastatic Colorectal Cancer
Brief Title: Nintedanib and Capecitabine in Treating Patients With Refractory Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Boehringer Ingelheim (Industry); National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 265514; NCI-2015-00223 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 265514 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH)
Record Dates: First submitted 2015-03-13; First posted 2015-03-19 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Colon Adenocarcinoma; Rectal Adenocarcinoma; Recurrent Colon Carcinoma; Recurrent Rectal Carcinoma; Stage IVA Colon Cancer; Stage IVA Rectal Cancer; Stage IVB Colon Cancer; Stage IVB Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Capecitabine; nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (capecitabine, nintedanib) (Experimental): Patients received capecitabine PO BID (every 12 hours) on days 1-14 and nintedanib PO BID (every 12 hours) on days 1-21. Courses repeated every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Capecitabine; Other: Laboratory Biomarker Analysis; Drug: Nintedanib; Other: Pharmacological Study
- Treatment (capecitabine , nintendanib) (Experimental): Patients receive the highest safe dose of the combination of nintedanib and capcitabine.
  Interventions: Drug: Nintedanib

INTERVENTIONS:
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
  Arms: Treatment (capecitabine, nintedanib)
Other: Laboratory Biomarker Analysis — Correlative studies
  Arms: Treatment (capecitabine, nintedanib)
Drug: Nintedanib — Given PO
  Other Names: BIBF 1120; BIBF-1120; Intedanib; Multitargeted Tyrosine Kinase Inhibitor BIBF 1120; tyrosine kinase inhibitor BIBF 1120; Vargatef
Other: Pharmacological Study — Correlative studies
  Arms: Treatment (capecitabine, nintedanib)

SUMMARY:
This phase I/II trial studies the side effects and best dose of nintedanib when given together with capecitabine and to see how well they work in treating patients with colorectal cancer that has not responded to previous treatment (refractory) and has spread to other places in the body (metastatic). Nintedanib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It may also block the growth of new blood vessels necessary for tumor growth. Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving nintedanib with capecitabine may be a better treatment for colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

* I. To estimate the maximum tolerated dose (MTD) and examine the dose-limiting toxicities of nintedanib when administered with capecitabine within the study population and, establish the recommended phase II dose (RP2D). (Phase I)
* II. To assess progression free survival at 18 weeks. (Phase II)

SECONDARY OBJECTIVES:

* I. To assess median progression free survival. (Phase II)
* II. To assess median overall survival from the date of enrollment to the time of death will be documented. (Phase II)
* III. To assess the objective response rate as measured by Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. (Phase II)
* IV. To assess the toxicity of dose regimen using the Cancer Therapy Evaluation Program (CTEP) National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE version 4.0). (Phase II)

TERTIARY OBJECTIVES:

* I. Measurement of circulating angiogenic cytokines (CAFs): vascular endothelial growth factor (VEGF), soluble vascular endothelial growth factor receptor (sVEGFR) 1/2, placental growth factor (PlGF), granulocyte macrophage colony-stimulating factor (GMCSF), leptin, interleukin (IL)-1 alpha (a), IL-8, IL-6, fibroblast growth factor basic (FGFb), osteopontin and pentraxin-3. (Phase II)
* II. Measurement of drug levels and pharmacokinetic (PK)/pharmacodynamic (PD) modeling. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of nintedanib followed by a phase II study.

Patients receive capecitabine orally (PO) twice daily (BID) (every 12 hours) on days 1-14 and nintedanib PO BID (every 12 hours) on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 28 days until resolution or satisfactory stabilization of persistent drug-related toxicity, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Hemoglobin >= 9 g/dL
* Absolute neutrophil count >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Creatinine =< 1.5 upper limit of normal (ULN) AND creatinine clearance (CrCl) > 50 mL/min by Cockcroft-Gault equation
* Males = (140 -age (yrs) (body weight (kg)/(72) (serum creatinine) (mg/dL)
* Females = 0.85 * (140-age (yrs) (body weight (kg)/(72)(serum creatinine (mg/dL)
* Bilirubin < ULN
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 1.5 ULN if without liver metastases
* AST/ALT =< 2.5 x ULN if with liver metastases
* Coagulation parameters: international normalized ratio (INR) =< 2, prothrombin time (PT) and partial thromboplastin time (PTT) < 1.5 X institutional ULN
* Have measurable disease per RECIST 1.1 criteria
* Histologically or cytologically proven adenocarcinoma of the colon or rectum
* Prior progression following a fluoropyrimidine-based therapy and progression following or intolerance to irinotecan and oxaliplatin, as well as anti-epidermal growth factor receptor (EGFR) therapy (e.g., panitumumab or cetuximab) for rat sarcoma viral oncogene homolog (RAS) wild-type patients
* Ability to swallow and retain oral medication
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry and for three months following completion of therapy; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Prior treatment with nintedanib
* Prior treatment with regorafenib
* Major injuries or surgery within the 4 weeks prior to initiation of therapy with incomplete wound healing or planned surgery during the on-study treatment period
* Uncontrolled hypertension: systolic blood pressure >= 160, diastolic blood pressure >= 90
* Urine protein/creatinine ratio >= 1.0
* History of clinically significant hemorrhagic or thrombotic event within the past 6 months, not including uncomplicated catheter-associated venous thrombosis; patients on anti-coagulation are not permitted to be on any oral formulations (warfarin, rivaroxaban, dabigatran, etc.) due to concern for drug-drug interaction
* Unstable angina, symptomatic congestive heart failure or cardiac arrhythmia requiring anti-arrhythmic therapy (beta-blockers, calcium channel blockers and digoxin are allowed)
* History of cerebrovascular or myocardial ischemia within 6 months of initiation
* Known inherited predisposition to bleeding or thrombosis
* Known active or chronic hepatitis B or C or human immunodeficiency virus (HIV)
* Untreated brain metastases
* History of second primary malignancy diagnosed within 3 years prior to enrollment, excluding:

  * In-situ cervical carcinoma
  * Superficial bladder cancer
  * Non-melanoma skin cancer
  * Stage I breast cancer
  * Low grade (Gleason =< 6) localized prostate cancer
  * Any additional malignancy which has been in clinical remission for at least 1 year
* Pregnant or nursing female participants
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the participant an unsuitable candidate to receive study drug
* Received an investigational agent within 4 weeks prior to enrollment
* PHASE I: History of intolerance to capecitabine at doses =< 1000 mg/m^2 BID, as defined by documented >= grade 3 hand-foot syndrome, documented severe diarrhea requiring hospitalization, or other documented severe adverse events (AEs) attributable to capecitabine
* PHASE II: History of intolerance to capecitabine at doses below 1000 mg/m^2 BID, as defined by documented >= grade 3 hand-foot syndrome; documented severe diarrhea requiring hospitalization; or other documented severe AEs attributable to capecitabine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-05-08 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2021-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christos Fountzilas, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Roswell Park Cancer Institute, Buffalo, New York

REFERENCES:
- [Derived] Boland PM, Ebos JML, Attwood K, Mastri M, Fountzilas C, Iyer RV, Banker C, Goey AKL, Bies R, Ma WW, Fakih M. A phase I/II study of nintedanib and capecitabine for refractory metastatic colorectal cancer. JNCI Cancer Spectr. 2024 Apr 30;8(3):pkae017. doi: 10.1093/jncics/pkae017. PMID 38697618

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: Capecitabine at 2000 mg/2, Nintedanib at 150 mg: Dose Level (Arm) 1: Capecitabine at 2000 mg/m2 PO daily and Nintedanib at 150 mg PO bid
  Capecitabine at 2000 mg/m2 will be administration will be twice daily for two weeks (the first 2 weeks of each 21 day cycle), followed by a 1 week rest. Nintedanib 150 mg will be administered twice daily for 21 days (i.e., 1 complete 3-week cycle). Both capecitabine and nintedanib may be taken together, with water, within 30 minutes following a meal. Doses should be separated by approximately 12 hours, with the PM dose being 12 hours (+/- 2 hours) after the AM dose.
- Dose Level 2: Capecitabine at 2000 mg/m2, Nintedanib at 200 mg: Dose Level (Arm) 2: Capecitabine at 2000 mg/m2 PO daily and Nintedanib at 200 mg PO bid
  Capecitabine at 2000 mg/m2 will be administration will be twice daily for two weeks (the first 2 weeks of each 21 day cycle), followed by a 1 week rest. Nintedanib 2000 mg will be administered twice daily for 21 days (i.e., 1 complete 3-week cycle). Both capecitabine and nintedanib may be taken together, with water, within 30 minutes following a meal. Doses should be separated by approximately 12 hours, with the PM dose being 12 hours (+/- 2 hours) after the AM dose.
Period: Overall Study
Arm/Group | Dose Level 1: Capecitabine at 2000 mg/2, Nintedanib at 150 mg | Dose Level 2: Capecitabine at 2000 mg/m2, Nintedanib at 200 mg
Started | 3 | 39
Completed | 3 | 32
Not Completed | 0 | 7
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Groups:
- Dose Level 1: Capecitabine at 2000 mg/m2, Nintedanib at 150 mg: Dose Level (Arm) 1: Capecitabine at 2000 mg/m2 PO daily and Nintedanib at 150 mg PO bid
  Capecitabine at 2000 mg/m2 will be administration will be twice daily for two weeks (the first 2 weeks of each 21 day cycle), followed by a 1 week rest. Nintedanib 150 mg will be administered twice daily for 21 days (i.e., 1 complete 3-week cycle). Both capecitabine and nintedanib may be taken together, with water, within 30 minutes following a meal. Doses should be separated by approximately 12 hours, with the PM dose being 12 hours (+/- 2 hours) after the AM dose.
- Dose Level 2: Capecitabine at 2000 mg/m2,Nintedanib at 200 mg: Dose Level (Arm) 2: Capecitabine at 2000 mg/m2 PO daily and Nintedanib at 200 mg PO bid
  Capecitabine at 2000 mg/m2 will be administration will be twice daily for two weeks (the first 2 weeks of each 21 day cycle), followed by a 1 week rest. Nintedanib 2000 mg will be administered twice daily for 21 days (i.e., 1 complete 3-week cycle). Both capecitabine and nintedanib may be taken together, with water, within 30 minutes following a meal. Doses should be separated by approximately 12 hours, with the PM dose being 12 hours (+/- 2 hours) after the AM dose.
- Total: Total of all reporting groups
Arm/Group | Dose Level 1: Capecitabine at 2000 mg/m2, Nintedanib at 150 mg | Dose Level 2: Capecitabine at 2000 mg/m2,Nintedanib at 200 mg | Total
Number analyzed (Participants) | 3 | 39 | 42
Age, Continuous [Mean (Full Range); unit: years] | 61.0 [55 to 63] | 57.3 [35 to 77] | 57.6 [35 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 22 | 24
  Male | 1 | 17 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 5 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 30 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
ECOG Status at Baseline [Count of Participants; unit: Participants] — ECOG Performance Status, Developed by the Eastern Cooperative Oncology Group, Robert L. Comis, MD
  GRADE
  0. Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    Grade 0 | 2 | 21 | 23
    Grade 1 | 1 | 18 | 19
Body Weight [Mean (Full Range); unit: Kilograms (kg)] | 69.2 [57.6 to 90.4] | 77.8 [41.1 to 126] | 77.2 [41.1 to 126]
Presence of liver metastasis [Count of Participants; unit: Participants] | 3 | 20 | 23

OUTCOME MEASURES:

1. Primary Outcome: To Examine the DLT
Description: The recommended Phase II dose is of the Nintedanib and Capecitabine combination is defined as the dose level that causes dose limiting toxicities (DLTs) in ≤ 1 out of 6 patients at highest dose level below the maximally administered dose.
  Capecitabine is fixed dose at 2000 mg/m2; while Nintedanib is evaluated at 150mg (dose level 1) and 200 mg (dose level 2).
Time Frame: At least 21 days.
Population: Patients who were evaluable for DLTs
Measure: Number; unit: mg
Groups:
- Treatment (Capecitabine, Nintedanib): Patients receive capecitabine PO BID (every 12 hours) on days 1-14 and nintedanib PO BID (every 12 hours) on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Capecitabine: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Nintedanib: Given PO
  Pharmacological Study: Correlative studies
Arm/Group | Treatment (Capecitabine, Nintedanib)
Number analyzed (Participants) | 9
mg | 200

2. Primary Outcome: Progression Free Survival (PFS) Rate, Defined as the Proportion of Patients Who Survive Without Disease Progression Via the RECIST Version 1.1 (Phase II)
Description: Progressive disease is defined as at least a 20% increase in the sum of diameters of target lesions (the sum must also demonstrate an absolute increase of at least 5 mm) or the appearance of new lesions.
  Will be summarized using standard Kaplan-Meier methods.
Time Frame: At 18 weeks
Population: All treated and eligible patients at dose level 2
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Capecitabine, Nintedanib)
Number analyzed (Participants) | 36
percentage of participants | 41.7 [29.2 to 55.3]

3. Secondary Outcome: Median PFS (Phase II)
Description: Progressive disease is defined as at least a 20% increase in the sum of diameters of target lesions (the sum must also demonstrate an absolute increase of at least 5 mm) or the appearance of new lesions. Estimates of median PFS will be obtained with corresponding 90% confidence intervals.
Time Frame: Up to 2 years
Population: All treated and eligible patients at dose level 2
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Capecitabine, Nintedanib)
Number analyzed (Participants) | 36
months | 3.4 [2.1 to 4.2]

4. Secondary Outcome: Median OS (Phase II)
Description: Overall survival is defined as time from date of subject enrollment to the date of death due to any cause. Estimates of median OS will be obtained with corresponding 90% confidence intervals.
Time Frame: From the date of enrollment to the time of death, assessed up to 2 years
Population: All treated and eligible patients at dose level 2
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Capecitabine, Nintedanib)
Number analyzed (Participants) | 36
months | 8.9 [5.9 to 13.8]

5. Secondary Outcome: Objective Response Rate
Description: Overall Response is defined as Complete Response: Disappearance of all target lesions and any lymph nodes must have a reduction in short axis to < 10 mm; or Partial Response: At least a 30% decrease in the sum of diameters of target lesions; or Stable Disease: Neither sufficient shrinkage to qualify for partial response, nor sufficient increase to qualify for progressive disease.
Time Frame: After every 3 cycles (9 weeks) of therapy.
Population: All treated and eligible patients at dose level 2
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Capecitabine, Nintedanib)
Number analyzed (Participants) | 36
percentage of participants | 58.3 [44.7 to 70.8]

6. Secondary Outcome: Aggregate Rates of Adverse Events Measured by CTCAE Version 4.0 (Phase II)
Description: Number of Participants with Adverse Events, Graded According to the CTEP NCI Common Terminology Criteria for Adverse Events (CTCAE Version 4.0).
Time Frame: Up to 30 days after the last dose of study drug
Population: All treated and eligible patients at dose level 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Capecitabine, Nintedanib)
Number analyzed (Participants) | 36
Participants
  Grade 1 | 3
  Grade 2 | 13
  Grade 3 | 16
  Grade 4 | 1
  Grade 5 | 3

ADVERSE EVENTS:
Time Frame: Day 1 of all Cycles, Cycle 1 Day 8 and Cycle 2 Day 8 (for phase 1 only), End of Treatment, an average of 102 days
Description: All treated and eligible patients
Arm/Group | Dose Level 1: Capecitabine at 2000 mg/m2, Nintedanib at 150 mg | Dose Level 2: Capecitabine at 2000 mg/m2,Nintedanib at 200 mg
All-Cause Mortality (participants affected / at risk) | 3/3 | 32/39
Serious Adverse Events (participants affected / at risk) | 0/3 | 10/39
Other Adverse Events (participants affected / at risk) | 3/3 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1: Capecitabine at 2000 mg/m2, Nintedanib at 150 mg (N=3) | Dose Level 2: Capecitabine at 2000 mg/m2,Nintedanib at 200 mg (N=39)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1: Capecitabine at 2000 mg/m2, Nintedanib at 150 mg (N=3) | Dose Level 2: Capecitabine at 2000 mg/m2,Nintedanib at 200 mg (N=39)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 14 (25)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 5 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 2 (2)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 2 (2)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 5 (6)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 10 (10)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (3)
Ascites (Gastrointestinal disorders) | 1 (1) | 2 (2)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 11 (14)
Diarrhoea (Gastrointestinal disorders) | 2 (4) | 22 (49)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 3 (3)
Flatulence (Gastrointestinal disorders) | 1 (1) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (6) | 27 (45)
Oral pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (7) | 5 (5)
Vomiting (Gastrointestinal disorders) | 3 (3) | 26 (45)
Asthenia (General disorders) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 3 (3)
Fatigue (General disorders) | 3 (4) | 23 (48)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Medical device pain (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 2 (4)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (2)
Oedema (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (2) | 6 (6)
Swelling (General disorders) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 3 (6)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Legionella infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (3)
Urinary tract infection (Infections and infestations) | 1 (2) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 16 (23)
Aspartate aminotransferase (Investigations) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 3 (4) | 19 (31)
Blood albumin decreased (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 16 (25)
Blood bilirubin increased (Investigations) | 0 (0) | 10 (16)
Blood creatinine increased (Investigations) | 0 (0) | 1 (5)
Blood sodium decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 2 (3)
Serum ferritin decreased (Investigations) | 0 (0) | 1 (1)
Transferrin saturation decreased (Investigations) | 0 (0) | 1 (1)
Urine protein, quantitative (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 7 (10)
White blood cell count decreased (Investigations) | 0 (0) | 5 (7)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 16 (27)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 11 (25)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (9)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 10 (13)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (4)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Bone marrow leukaemic cell infiltration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 8 (8)
Dysarthria (Nervous system disorders) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 8 (9)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 9 (10)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Taste disorder (Nervous system disorders) | 0 (0) | 4 (4)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Catatonia (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (7)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (3)
Renal injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 8 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 8 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 8 (9)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (11) | 15 (36)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 3 (3)
Hot flush (Vascular disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 2 (7) | 9 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-16): https://cdn.clinicaltrials.gov/large-docs/55/NCT02393755/Prot_SAP_000.pdf